CLINICAL TRIAL: NCT05302700
Title: The Effectiveness of Early Parental Sensitivity Intervention on Attachment, Parenting Confidence and Parental Stress of Preterm Infant Mothers
Brief Title: Effectiveness of Early Parental Sensitivity Intervention for Preterm Infant Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Y_110_0501
Record Dates: First submitted 2022-03-15; First posted 2022-03-31 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-03

CONDITIONS: Attachment; Parental Stress
Keywords: preterm infant mothers; early; parental sensitivity intervention; attachment; parenting confidence; parental stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Parental Sensitivity Intervention Program (Experimental): The protocol will last five to seven days for preterm infant mothers.
  Interventions: Behavioral: Early Parental Sensitivity Intervention
- Control group (No Intervention): The control group received general routine nursing guidance.

INTERVENTIONS:
Behavioral: Early Parental Sensitivity Intervention — Parental sensitivity intervention include (1)Establish an emotional connection：Using the VR tour to introduce the environment, instruments and equipment of the neonatal intensive care unit, appearance of premature infants and pipeline wires on their bodies .(2)maintain physical proximity:proactively provide mothers with the opportunity to touch the body of preterm infants.(3) parents must understand their infant's cues:Using the Premature Infant Behavioral Clues Teaching Materials to play video and we will discuss and respond to the mother's questions.(4)engage in his/her care and communicate appropriately with him/her:We will discuss the behavioral clues of the preterm infant with the mother next to the incubator, encourage the mother to ask questions and participate in care activities such as changing diapers and stamping the baby's footprints on the card, asking the mother to write down the number of days of birth, corrected age, weight and what she wants to say for her baby.
  Arms: Early Parental Sensitivity Intervention Program

SUMMARY:
In Taiwan, according to the birth notification statistics of the Ministry of Health and Welfare. 164,496 newborns were born in 2020, with preterm births accounting for about 11.58%.Most preterm infants need to be hospitalized for highly specialized care, resulting in the separation of preterm infants from their parents after birth, which may have a negative impact on the healthy attachment development between parents and preterm infants. Moreover, due to the vulnerability of preterm infants, parents often lack the confidence to take care of them.

DETAILED DESCRIPTION:
The study was a quantitative study of a randomized controlled trial, designed by experimental research method. Using GPower 3.1.2 to estimate the number of samples, and the statistical method chosen was Repeated measures ANOVA, the sample size was 80.

The subjects were divided into two groups, The control group received general routine nursing guidance, while the experimental group received general routine nursing guidance and early parental sensitivity intervention program. Using the NICU VR Tour and Premature Infant Behavioral Clues Teaching Materials as educational tools for early parental sensitivity intervention program. The outcome used the Maternal Attachment Inventory, Maternal Confidence Questionnaire and Parental Stressor Scale: Infant Hospitalization as evaluated tools.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants:

   1. Preterm infants less than 37 weeks gestation and hospitalized in the NICU
   2. The birth weight is classified as VLBW and LBW, and the birth weight is between 1,000-2,499gm
2. Preterm infant mothers:

   1. Children have not been hospitalized in the NICU in the past
   2. At least 20 years old
   3. They can speak Chinese, Taiwanese fluently and need to be literate

Exclusion Criteria:

1. Preterm infants :

   1. Combined congenital diseases and chromosomal abnormalities
   2. Immediate surgery, first aid and unstable vital signs are necessary after birth
   3. The birth weight is classified as ELBW, and the birth weight is less than 1,000gm
2. Preterm infant mothers:

   1. Hospitalized in the intensive care unit

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Maternal Attachment Inventory | On the fifth to seventh day after birth of preterm infant.
  Using the Maternal Attachment Inventory to measure mother-infant attachment.There are 22 items on the scale,each item was scored using a 4-point Likert scale.The total score ranges from 22 to 88, with higher scores indicating better attachment.
Maternal Confidence Questionnaire | On the fifth to seventh day after birth of preterm infant.
  Using the Maternal Confidence Questionnaire to measure parenting confidence.There are 14 items on the scale,each item was scored using a 5-point Likert scale.The total score ranges from 14 to 70, with higher scores indicating better parenting confidence.
Parental Stressor Scale: Infant Hospitalization | On the fifth to seventh day after birth of preterm infant.
  Using the Parental Stressor Scale: Infant Hospitalization to measure parental stress.There are 21 items on the scale,each item was scored using a 5-point Likert scale.The total score ranges from 21 to 105, with higher scores indicating greater stress.

SECONDARY OUTCOMES:
Maternal Attachment Inventory | The first month of birth of preterm infant.
  Using the Maternal Attachment Inventory to measure mother-infant attachment.There are 22 items on the scale,each item was scored using a 4-point Likert scale.The total score ranges from 22 to 88, with higher scores indicating better attachment.
Maternal Confidence Questionnaire | The first month of birth of preterm infant.
  Using the Maternal Confidence Questionnaire to measure parenting confidence.There are 14 items on the scale,each item was scored using a 5-point Likert scale.The total score ranges from 14 to 70, with higher scores indicating better parenting confidence.
Parental Stressor Scale: Infant Hospitalization | The first month of birth of preterm infant.
  Using the Parental Stressor Scale: Infant Hospitalization to measure parental stress.There are 21 items on the scale,each item was scored using a 5-point Likert scale.The total score ranges from 21 to 105, with higher scores indicating greater stress.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavallee A, Aita M, Bourbonnais A, De Clifford-Faugere G. Effectiveness of early interventions for parental sensitivity following preterm birth: a systematic review protocol. Syst Rev. 2017 Mar 23;6(1):62. doi: 10.1186/s13643-017-0459-x. PMID 28335806
- [Background] Dunham MM, Marin T. NICU Maternal-Infant Bonding: Virtual Visitation as a Bonding Enhancement Tool. J Perinat Neonatal Nurs. 2020 Apr/Jun;34(2):171-177. doi: 10.1097/JPN.0000000000000484. PMID 32332447
- [Background] Ioannou A, Papastavrou E, Avraamides MN, Charalambous A. Virtual Reality and Symptoms Management of Anxiety, Depression, Fatigue, and Pain: A Systematic Review. SAGE Open Nurs. 2020 Aug 27;6:2377960820936163. doi: 10.1177/2377960820936163. eCollection 2020 Jan-Dec. PMID 33415290
- [Background] Kim AR, Kim SY, Yun JE. Attachment and relationship-based interventions for families during neonatal intensive care hospitalization: a study protocol for a systematic review and meta-analysis. Syst Rev. 2020 Mar 21;9(1):61. doi: 10.1186/s13643-020-01331-8. PMID 32199458